CLINICAL TRIAL: NCT00660595
Title: A Pilot Study of Three-Week, Randomised, Open Comparison in Schizophrenic In-patients Treated With Quetiapine Prolong or Oral Risperidone at Flexible Dose
Brief Title: Study in Schizophrenic In-patients Treated With Quetiapine Prolong or Oral Risperidone at Flexible Dose
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: To difficult to recruit patients in the acute setting
Sponsor: AstraZeneca (Industry)
Responsible Party: Hans Eriksson - Medical Science Director, AstraZeneca
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D1443L00042
Record Dates: First submitted 2008-04-14; First posted 2008-04-17 (Estimated); Results first posted 2010-09-17 (Estimated); Last update posted 2010-09-17 (Estimated); Status verified 2010-08

CONDITIONS: Schizophrenic Disorders
Keywords: Schizophrenia; Schizoaffective psychosis; Schizophreniformic psychosis; Pilot study; Quetiapine Prolong; Risperidone
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders | interventions — Quetiapine Fumarate; Risperidone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Oral
  Interventions: Drug: Quetiapine
- 2 (Active Comparator): Oral
  Interventions: Drug: Risperidone

INTERVENTIONS:
Drug: Quetiapine — Oral administration
  Other Names: Seroquel
  Arms: 1
Drug: Risperidone — Oral administration
  Other Names: Risperdal
  Arms: 2

SUMMARY:
This pilot trial in Finland is designed to evaluate in a randomized fashion change of agitation in acute schizophrenic patients (Schizophrenia or Schizoaffective psychosis or Schizophreniformic psychosis)Diagnostic and Statistical Manual (DSM - IV) with the first visits on days 1, 2, 4 or 5 and 7 ± 1.

ELIGIBILITY:
Inclusion Criteria:

* In the opinion of the Investigator, requirement for treatment for an acute episode of schizophrenia, schizoaffective disorder or schizophreniformic psychosis (according to DSM-IV diagnostic criteria), Positive and Negative Symptoms Scale (PANSS) ≥ 65, CGI ≥ 4

Exclusion Criteria:

* Pregnancy or lactation
* In-patients/hospitalized > 7 days before enrollment
* Known intolerance or lack of response to quetiapine fumarate or risperidone, as judged by the investigator

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2008-09; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yrjö Ovaskainen, MD, Study Director — AstraZeneca Finland; Hannu Koponen, MD, PhD, Principal Investigator — Kuopio University
Locations (4):
- Finland (4):
  - Research Site, Harjavalta
  - Research Site, Helsinki
  - Research Site, Pitkäniemi
  - Research Site, Turku

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Two recruiting sites between 13 may 2008 and 28 Jan 2009: Aurora Hospital Helsinki and Pitkäniemi Hospital Tampere.
Pre-assignment Details: Site 01 pre-screened 19 subjects, two were randomised, 12 did not consent to participate and five were not included due to other reasons.One subject completed the study and the other discontinued from the study on Day 2 (subject escaped from the hospital).Site 03 pre-screened 10 subjects, of which only one completed the study.
Groups:
- Seroquel: Quetiapine Prolong, oral administration
- Risperdal: Risperidone, oral administration
Period: Overall Study
Arm/Group | Seroquel | Risperdal
Started | 19 | 10
Completed | 1 | 1 (One of the two was lost to follow-up)
Not Completed | 18 | 9
Not completed — Lost to Follow-up | 0 | 1
Not completed — Did not consent to participate in study | 12 | 8
Not completed — Participant left hospital | 1 | 0
Not completed — Non Specified reasons | 5 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Seroquel | Risperdal | Total
Number analyzed (Participants) | 19 | 10 | 29
Age Continuous [Mean (Full Range); unit: years] | 47 [47 to 47] | 51 [39 to 63] | 49 [47 to 63]
Gender [Number; unit: Participants] — randomised participants
  Participants
    Female | 1 | 1 | 2
    Male | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Positive and Negative Symptoms Scale, Excitatory Subscale (PANSS-EC) Score (Time Frame: 3 Weeks)
Description: PANSS-EC score change was to be measured by calculating the difference between baseline score and 3 week's score. The PANSS-EC consists of 5 items (Poor IMpulse Control, Tension, Hostility, Uncooperativeness, and Excitement), each with associated descriptors. Each descriptor is rated on a 7 point scale from 1 = (absence of any symptom) to 7 = (extremely severe symptoms).
Time Frame: baseline and 3 weeks
Measure: Number; unit: units on a scale
Arm/Group | Seroquel | Risperdal
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Change From Baseline in Clinical Global Impression, Severity Scale (CGI-S) and in Absolute Clinical Global Impression, Improvement Scale (CGI-I) (Performed 4 Times/ 3 Weeks)
Description: The CGI change was to be measured by calculating the difference between baseline score and 3 week's score. CGI-S Score of 1 = no illness to score of 7 = extremely ill. CGI-I Score of 1 =very much improved since the initiation of treatment to 7=very much worse since the initiation of treatment
Time Frame: baseline and 3 weeks
Measure: Number; unit: units on a scale
Arm/Group | Seroquel | Risperdal
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Change From Baseline in Overt Aggression Scale (OAS) (Performed 6 Times/ 3 Weeks)
Description: The Overt Agression Scale (OAS) change was to be measured by calculating the difference between baseline score and 3 week's score. Score between 1 and 16 verbal aggression (OAS 1, score 1-4), physical aggression against objects (OAS 2, score 5-8), physical aggression against self (OAS 3, score 9-11) and physical aggression against other people (OAS 4, score 12-16).
Time Frame: baseline and 3 weeks
Measure: Number; unit: units on a scale
Arm/Group | Seroquel | Risperdal
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Change From Baseline in Total Positive and Negative Symptoms Scale (PANSS Score) (Performed 5 Times/ 3 Weeks)
Description: PANSS score change was to be measured by calculating the difference between baseline score and 3 week's score. The PANSS consists of 7 positive and 11 negative items each with associated descriptors. Each descriptor is rated on a 7 point scale from 1=(absence of any symptom) to 7=(extremely severe symptoms).
Time Frame: baseline and 3 weeks
Measure: Number; unit: units on a scale
Arm/Group | Seroquel | Risperdal
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | Seroquel | Risperdal
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/1
Other Adverse Events (participants affected / at risk) | 0/1 | 1/1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Seroquel (N=1) | Risperdal (N=1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1
Elevated Prolactin Level (Endocrine disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less